CLINICAL TRIAL: NCT01361087
Title: Circulating Transforming Growth Factor Beta (TGF-β) in Individuals With
Brief Title: Circulating Transforming Growth Factor Beta (TGF-β) in Individuals With Marfan Syndrome
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No outside recruitment of subjects from Main Atenolol VS Losartan NIH study
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB # 2011-14507
Record Dates: First submitted 2011-05-25; First posted 2011-05-26 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Marfan Syndrome
Keywords: TGF-B blood levels Atenolol vs, Losartan Study, NIH, NIHLB and NMF
MeSH Terms: conditions — Marfan Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood draw — This study includes one blood draw to measure circulating blood levels of TGF-B.

SUMMARY:
Transforming Growth Factor Beta (TGF-β) is a protein that controls proliferation, cellular differentiation, and other functions in most cells. TGF-β levels play a major role in the pathogenesis of Marfan syndrome, a disease characterized by disproportionate height, long extremities, lens dislocation in the eyes and heart complications such as mitral valve prolapse and aortic enlargement increasing the likelihood of aortic dissection. While the underlying defect in Marfan syndrome is faulty synthesis of the glycoprotein fibrillin I, normally an important component of elastic fibers it has been shown that the Marfan syndrome phenotype can be relieved by addition of a TGF-β antagonist in affected mice.

DETAILED DESCRIPTION:
Transforming Growth Factor Beta (TGF-β) is a protein that controls proliferation, cellular differentiation, and other functions in most cells. TGF-β levels play a major role in the pathogenesis of Marfan syndrome, a disease characterized by disproportionate height, long extremities, lens dislocation in the eyes and heart complications such as mitral valve prolapse and aortic enlargement increasing the likelihood of aortic dissection. While the underlying defect in Marfan syndrome is faulty synthesis of the glycoprotein fibrillin I, normally an important component of elastic fibers it has been shown that the Marfan syndrome phenotype can be relieved by addition of a TGF-β antagonist in affected mice. This suggest that while the symptoms of Marfan syndrome may seem consistent with a connective tissue disorder, the mechanism is more likely related to reduced sequestration of TGF-β by fibrillin.

ELIGIBILITY:
Inclusion Criteria:

* Individual with Marfan syndrome consented in to the Main Atenolol Vs. Losartan NIH study.

Exclusion Criteria:

* Subjects in the main PHN Marfan trial who have not achieved the maintenance drug dosing or who have stopped taking study drug.

Ages: 6 Months to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine if circulating levels of TGF-β correlate with treatment arms: Atenolol vs. Losartan. | 1 year

SECONDARY OUTCOMES:
To determine if circulating levels of TGF-β correlate with clinical outcomes within a treatment group or independent treatment groups. | 1 year
  These clinical outcomes may be a change in aortic root Z-score, final aortic root dimension, final aortic root Z-score and other clinical outcomes in the main Marfan trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Memorial Hospital Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided